CLINICAL TRIAL: NCT05836792
Title: The Effect of Cycle Ergometer With Biofeedback on Deep Sensation in Elderly Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nilay Aral (Other)
Collaborators: Sante Medical Center (Other)
Responsible Party: Sponsor-Investigator, Nilay Aral, Physiotherapist, Yeditepe University
Organization: Yeditepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20203034001
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Knee Osteoarthritis; Sensation Disorders
Keywords: Knee Osteoarthritis; Deep Sensation; Cycle Ergometer; Biofeedback
MeSH Terms: conditions — Osteoarthritis, Knee; Sensation Disorders | interventions — Transcutaneous Electric Nerve Stimulation; Ultrasonography; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycle Ergometer Group (CEG) (Experimental): Isometric exercises Transcutaneous electrical nerve stimulation Ultrasound Cycle ergometer
  Interventions: Other: Cycle Ergometer; Device: Transcutaneous electrical nerve stimulation; Device: Ultrasound; Other: Isometric exercises
- Control Group (Active Comparator): Isometric exercises Transcutaneous electrical nerve stimulation Ultrasound
  Interventions: Device: Transcutaneous electrical nerve stimulation; Device: Ultrasound; Other: Isometric exercises

INTERVENTIONS:
Other: Cycle Ergometer — Patients will attend cycle ergometer exercise. Volunteers will monitor their pedaling forces as right and left force. They will try to make these forces equal while they are pedaling.
  Arms: Cycle Ergometer Group (CEG)
Device: Transcutaneous electrical nerve stimulation — Transcutaneous electrical nerve stimulation will be used for the reduction of pain. TENS will be used 5 times in a week for 3 weeks. Each procedure will take 20 minutes.
  Other Names: TENS
Device: Ultrasound — Ultrasound will be used for increase the permeability of cells to treat pain and inflammation. US will be used 5 times in a week for 3 weeks. Each procedure will take 5 minutes
  Other Names: US
Other: Isometric exercises — The aim of the isometric exercises is increasing muscle strength. Each session patients will do quadriceps isometric exercises 5 times in a week for 3 weeks

SUMMARY:
The aim of the randomized controlled study is to investigate the effects of the cycle ergometer with biofeedback on deep sensation in elderly people who has knee osteoarthritis

DETAILED DESCRIPTION:
Participants will be randomly divided and registered into 2 groups: Thera-train tigo group (TG) or control group(CP)

For 20 participants 20 minute tens, 5 minute ultrasound, 10 times with 2 sets quadriceps isometric exercise will be applied. The other 20 participants will use Thera-train tigo for 20 minute in addition to tens, us, quadriceps isometric exercise.

Conditions of the participants will be measured before(1st day) and after(15th day) a span of 3 week treatment. We will use Demographic Information Questionnaire, Western Ontario and McMaster Universities (WOMAC) osteoarthritis index, Physical Activity Scale for the Eldery (PASE) and 6 minute walking test for all patients. Then we will measure knee vibration sense with diapason. Knee joint position sense will be measured with a digital goniometer.

ELIGIBILITY:
Inclusion Criteria:

Knee osteoarthritis (Kellgren-Lawrance score between 1-3)

Exclusion Criteria:

* Previous knee surgery
* Diabetus Mellitus
* Thyroid disease
* Visual deficit
* Gait disorder
* Mental Disability
* Presence of neuropathy

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Diapason survey | 3 weeks
  Diapason will be used to survey vibration sense to evaluate deep sensation
Digital Goniometer | 3 weeks
  Digital Goniometer will be used to measure angle of the knee position to evaluate deep sensation.
6 Minute Walking Test (6MWT) | 3 weeks
  Six Minute walking test will be used to evaluate functional capacity of volunteers

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 3 weeks
  WOMAC is a patient-reported outcome measure for the assessment of lower limb osteoarthritis
Physical Activity Scale for the Elderly (PASE) | 3 weeks
  Physical Activity Scale for the Elderly (PASE) will be used to evaluate the physical activities of individuals. Higher scores show the higher physical activity level.

CONTACTS AND LOCATIONS:
Locations (1):
- Sante Medical Center, Istanbul, Kadıköy, Turkey (Türkiye)